CLINICAL TRIAL: NCT06673316
Title: Integrating Design Thinking Into Undergraduate Nursing Education: a Pilot RCT
Brief Title: Integrating Design Thinking Into Undergraduate Nursing Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Carmen Chan Yip Wing-han, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-0219; SBRE-24-0219 (Other: Survey and Behavioural Research Ethics)
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Nurse Training
Keywords: Design thinking; Nursing education; Problem-solving skills; Empathy; Creativity; Patient-centered care attitude; Collaboration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants in the experimental group will receive a 3-hour design thinking workshop. The workshop will cover the five stages of design thinking, allowing students to apply these principles to real-world healthcare challenges in their future practice
  Interventions: Other: Design thinking workshop
- Control group (No Intervention): will NOT receive design thinking workshop

INTERVENTIONS:
Other: Design thinking workshop — The workshop will cover the five stages of design thinking, allowing students to apply these principles to real-world healthcare challenges in their future practice.
  Arms: Intervention group

SUMMARY:
Previous studies have demonstrated that design thinking workshops can indeed produce these effects in healthcare education settings. However, its effectiveness in nursing curriculum is inconclusive. This research project aims to introduce and integrate design thinking principles into the undergraduate nursing program at the Chinese University of Hong Kong (CUHK), the Nethersole School of Nursing. By implementing a comprehensive study encompassing desktop research, a 3-hour introductory workshop, and pre- and post-evaluations over a 9-month period, the investigators seek to enhance nursing students' problem-solving skills, empathy, creativity, collaboration, and patient-centered care attitude.

DETAILED DESCRIPTION:
Subjects A group of 50 second-year undergraduate nursing students at CUHK Nethersole School of Nursing who volunteer to participate in the research. Participants will be randomly assigned to either: i) Intervention group (n=25): Receives the design thinking workshop; ii) Control group (n=25): Receives no intervention (continues with regular curriculum). According to Hertzog (2008), a minimum of 25 subjects per group would be considered sufficient for the purposes of pilot testing. Students who have prior experience in joining design thinking workshop will be excluded.

Methodology This study employs a pilot randomized controlled design to evaluate the impact of a design thinking workshop on undergraduate nursing students' problem-solving abilities and related skills. The methodology encompasses a comprehensive literature review, pre- and post-workshop assessments, and a 3-hour introductory workshop on design thinking principles applied to healthcare challenges.

1. Systematic review and preparation of material A systematic review will be conducted to examine existing applications of design thinking in healthcare education, particularly in nursing, informing workshop curriculum development in terms of content, delivery method and evaluation approach.
2. Pre-Workshop Evaluation An online survey one month before the workshop will be conducted to assess participants' baseline skills and attitudes using validated instruments. These instruments measure problem-solving abilities, empathy, creativity, collaboration, and patient-centered care attitudes.
3. Design Thinking Workshop A 3-hour introductory workshop will cover the five stages of design thinking: Empathize, Define, Ideate, Prototype, and Test. Students will work on scenario of real-world healthcare challenges, and apply design thinking principles to develop innovative solutions.
4. Post-Workshop Evaluation Immediately after the workshop, participants will complete a post-workshop survey using the same instruments as the pre-workshop evaluation, allowing for comparison of scores.

ELIGIBILITY:
Inclusion Criteria:

- Undergraduate nursing students at CUHK Nethersole School of Nursing who volunteer to participate in the research.

Exclusion Criteria:

* Nil

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Problem-solving Abilities | Baseline
  rating on the Eight subscales of capabilities in Student engagement questionnaire (SEQ) (1=Strongly disagree, 5= Strongly Agree)
Problem-solving Abilities | immediately after workshop
  rating on the Eight subscales of capabilities in Student engagement questionnaire (SEQ) (1=Strongly disagree, 5= Strongly Agree)

SECONDARY OUTCOMES:
Creativity | Baseline
  rating on the Eight subscales of capabilities in Student engagement questionnaire (SEQ) (1=Strongly disagree, 5= Strongly Agree)
Creativity | immediately after workshop
  rating on the Eight subscales of capabilities in Student engagement questionnaire (SEQ) (1=Strongly disagree, 5= Strongly Agree)
Collaboration | Baseline
  rating on the Eight subscales of capabilities in Student engagement questionnaire (SEQ) (1=Strongly disagree, 5= Strongly Agree)
Collaboration | immediately after workshop
  rating on the Eight subscales of capabilities in Student engagement questionnaire (SEQ) (1=Strongly disagree, 5= Strongly Agree)
Empathy | Baseline
  rating on the Jefferson Scale of Empathy - Health Professions Student Version (JSE-HPS) (1=Strongly disagree, 5= Strongly Agree)
Empathy | immediately after workshop
  rating on the Jefferson Scale of Empathy - Health Professions Student Version (JSE-HPS) (1=Strongly disagree, 5= Strongly Agree)
Patient-centered Care attitude | Baseline
  rating on the Patient-Practitioner Orientation Scale (PPOS), 1= strongly disagree, 5=strongly agree
Patient-centered Care attitude | immediately after workshop
  rating on the Patient-Practitioner Orientation Scale (PPOS), 1= strongly disagree, 5=strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Carmen WH Chan, Principal Investigator — The Nethersole School of Nursing
Locations (1):
- The Nethersole School of Nursing, Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No